CLINICAL TRIAL: NCT06766591
Title: Ivonescimab Combined With Chemotherapy for EGFR Mutant NSCLC With Leptomeningeal Metastasis After EGFR TKIs Resistance: A Multicenter Observational Study.
Brief Title: Ivonescimab Combined With Chemotherapy for the Treatment of Leptomeningeal Metastases Failed to EGFR-TKIs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Collaborators: Henan Cancer Hospital (Other Government); Three Gorges Hospital of Chongqing University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY110-01
Record Dates: First submitted 2024-12-22; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: NSCLC; Chemotherapy; Leptomeningeal Metastases; EGFR-TKI; AK112
Keywords: Ivonescimab; NSCLC; leptomeningeal metastases; EGFR-TKI; VEGF; PD-1/VEGF bispecific antibody
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivonescimab combined with chemotherapy (Experimental)
  Interventions: Drug: Ivonescimab combined with chemotherapy

INTERVENTIONS:
Drug: Ivonescimab combined with chemotherapy — Ivonescimab combined with chemotherapy. The specific chemotherapy regimen is based on the real world.

SUMMARY:
Research objective Main purpose Exploring the real-world effectiveness of Ivonescimab combined with chemotherapy for EGFR mutant NSCLC with leptomeningeal metastasis after EGFR-TKIs resistance. Outcome measure: Real world intracranial disease-free survival time (iPFS).

Secondary purpose Federation patterns: describing different treatment modes in the real world; Outcome measures: Combination chemotherapy regimen and duration of chemotherapy.

Efficacy: Further explore the effectiveness of Ivonescimab combined with chemotherapy for EGFR mutant NSCLC with leptomeningeal metastasis failed with EGFR-TKI treatment; Outcome measures: Objective response rate (LM-ORR), duration of intracranial response (iDoR), overall progression free survival (PFS), overall survival (OS), improvement in neurological function, CSF response rate based on CSF cytology.

Safety: Explore the safety of Ivonescimab combined with chemotherapy for NSCLC patients with leptomeningeal metastases who have failed EGFR-TKI treatment; Outcome measures: incidence of adverse events (TEAEs), laboratory test outliers, and serious adverse events (SAEs).

Research endpoint Primary endpoint

* iPFS (intracranial progression free survival). Secondary endpoint
* Efficacy: leptomeningeal ORR (LM-ORR), intracranial duration of response (iDoR), overall progression free survival (PFS), overall survival (OS), improvement in neurological function, and CSF response rate based on CSF cytology;
* Safety: Determine the incidence and severity of adverse events (AE) and serious adverse events (SAE) according to NCI-CTCAE5.0 standards; Changes in vital signs, laboratory abnormalities, and quality of life scores.

Exploratory endpoint: efficacy related biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-75y
* EGFR mutation NSCLC
* LM was diagnosed through head enhanced MRI or (and) CSF cytology
* EGFR activation mutations were positive
* Patients who have failed to first or second-generation EGFR-TKI treatment，without T790M mutation; or failed to third-generation EGFR-TKI treatment
* Hematological, coagulation, renal and liver function is sufficient
* Women of childbearing age must undergo a pregnancy test and the result must be negative

Exclusion Criteria:

* Patients with squamous cell carcinoma, large cell carcinoma, mixed cell lung cancer
* The patient has other driver genes that can be treated with targeted drugs
* Subjects who have previously received immunotherapy with a discontinuation time of less than 3 months
* Received EGFR-TKI treatment within one week prior to the first administration
* Received non-specific immunomodulatory therapy
* Clinical manifestations of neurological failure
* Non malignant neurological disorders
* Radiotherapy for the chest and whole brain should be completed within 4 weeks before enrollment
* Tumor surrounded important blood vessels or had obvious necrosis or cavities
* Tumor has invaded important surrounding organs and blood vessels
* History of severe bleeding tendency or coagulation dysfunction
* The risk of developing esophagotracheal fistula or esophageal pleural fistula

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
intracranial progression free survival(iPFS) | From enrollment to the end of treatment at 12 months
  Treatment initiation to intracranial progression/death/deadline for last follow-up

SECONDARY OUTCOMES:
PFS | From enrollment to the end of treatment at 12 months
  Treatment start to PD/death/deadline for last follow-up
OS | From enrollment to the end of treatment at 18 months
  The time from randomization to death (for any reason)
iDoR | From enrollment to the end of treatment at 12 months
  The time from the first assessment of intracranial lesions as CR or PR to the first assessment as PD or death from any cause

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheng WC, Wang G, Mei Q. Ivonescimab Plus Chemotherapy in Patients With EGFR Variant Non-Small Cell Lung Cancer. JAMA. 2025 Jan 14;333(2):172. doi: 10.1001/jama.2024.23088. No abstract available. PMID 39661367
- [Result] Liu Z, Shan D, Han X. Ivonescimab Plus Chemotherapy in Patients With EGFR Variant Non-Small Cell Lung Cancer. JAMA. 2025 Jan 14;333(2):172-173. doi: 10.1001/jama.2024.23091. No abstract available. PMID 39661345
- [Result] Fang W, Li W, Zhang L. Ivonescimab Plus Chemotherapy in Patients With EGFR Variant Non-Small Cell Lung Cancer-Reply. JAMA. 2025 Jan 14;333(2):173-174. doi: 10.1001/jama.2024.23094. No abstract available. PMID 39661384
- [Result] Frentzas S, Austria Mislang AR, Lemech C, Nagrial A, Underhill C, Wang W, Wang ZM, Li B, Xia Y, Coward JIG. Phase 1a dose escalation study of ivonescimab (AK112/SMT112), an anti-PD-1/VEGF-A bispecific antibody, in patients with advanced solid tumors. J Immunother Cancer. 2024 Apr 19;12(4):e008037. doi: 10.1136/jitc-2023-008037. PMID 38642937
- [Result] Dhillon S. Ivonescimab: First Approval. Drugs. 2024 Sep;84(9):1135-1142. doi: 10.1007/s40265-024-02073-w. Epub 2024 Jul 29. PMID 39073550
- [Result] HARMONi-A Study Investigators; Fang W, Zhao Y, Luo Y, Yang R, Huang Y, He Z, Zhao H, Li M, Li K, Song Q, Du X, Sun Y, Li W, Xu F, Wang Z, Yang K, Fan Y, Liu B, Zhao H, Hu Y, Jia L, Xu S, Yi T, Lv D, Lan H, Li M, Liang W, Wang Y, Yang H, Jia Y, Chen Y, Lu J, Feng J, Liu C, Zhou M, Zhou J, Liu X, Zhou N, He M, Dong X, Chen H, Chen Y, Su H, Li X, Zhang Z, Yang L, Cheng Y, Chen L, Hou X, Zhang Y, Guo J, Wang Z, Lu H, Wu D, Feng W, Li W, Huang J, Wang Y, Song X, Peng J, Liu L, Guo Y, Li W, Lu D, Hu M, Wang ZM, Li B, Xia M, Zhang L. Ivonescimab Plus Chemotherapy in Non-Small Cell Lung Cancer With EGFR Variant: A Randomized Clinical Trial. JAMA. 2024 Aug 20;332(7):561-570. doi: 10.1001/jama.2024.10613. PMID 38820549
- [Result] Wang L, Luo Y, Ren S, Zhang Z, Xiong A, Su C, Zhou J, Yu X, Hu Y, Zhang X, Dong X, Meng S, Wu F, Hou X, Dai Y, Song W, Li B, Wang ZM, Xia Y, Zhou C. A Phase 1b Study of Ivonescimab, a Programmed Cell Death Protein-1 and Vascular Endothelial Growth Factor Bispecific Antibody, as First- or Second-Line Therapy for Advanced or Metastatic Immunotherapy-Naive NSCLC. J Thorac Oncol. 2024 Mar;19(3):465-475. doi: 10.1016/j.jtho.2023.10.014. Epub 2023 Oct 23. PMID 37879536
- [Result] Voron T, Colussi O, Marcheteau E, Pernot S, Nizard M, Pointet AL, Latreche S, Bergaya S, Benhamouda N, Tanchot C, Stockmann C, Combe P, Berger A, Zinzindohoue F, Yagita H, Tartour E, Taieb J, Terme M. VEGF-A modulates expression of inhibitory checkpoints on CD8+ T cells in tumors. J Exp Med. 2015 Feb 9;212(2):139-48. doi: 10.1084/jem.20140559. Epub 2015 Jan 19. PMID 25601652